CLINICAL TRIAL: NCT05738395
Title: Typical and Atypical Symptoms of Frey's Syndrome: a Pilot Study
Brief Title: Symptoms of Frey's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Marchese Maria Raffaella, Medical Doctor, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3494
Record Dates: First submitted 2023-02-01; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Parotid Neoplasms
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questions — Questions

SUMMARY:
The goal of this observational study is to describe the prevalence of typical and atypical signs and symptoms of Frey's syndrome, the affected areas and the severity of each symptom/sign.

Participants will be asked will asked about

* Presence or the absence of: a. gustatory sweating; b. gustatory flushing; c. gustatory itching; d. paresthesia; e. pain
* Grade of severity: a. absence; b. mild; c. moderate; d. almost severe; e. severe
* Affected area: a. preauricular; b. retroauricolar; c. temporal; d. retrangulomandibular; e. cheek

DETAILED DESCRIPTION:
The Frey's syndrome classically appears with sweating and hyperemia that occur almost immediately after tasting foods, particularly spicy ones, in the distribution of the auriculotemporal nerve region hence it is also called "auriculotemporal syndrome". The synkinetic mechanism for Frey's syndrome supposes an aberrant regeneration of the parasympathetic fibers because they normally innervate the parotid gland and, after losing their parotid targets, they regenerate to innervate the facial skin vessels and sweat glands. As a consequence, this results in a local vasodilatation (gustatory flushing) and localized sweating (gustatory sweating) of the sympathetically void skin in response to mastication and salivation (Drummond PD, 2002; Rustemeyer J et al., 2008; Neumann A e al., 2011; Gardner WJ et al., 1956). The etiology may be traumatic (parotidectomy, abscess drainage, bullet wound) (Rouyer J., 1959; Botkin S., 1875) or nontraumatic (autonomic neuropathy in diabetes mellitus, herpes zoster infection, metabolic diseases, etc.) (New GB, 1922). The most frequent etiologic factor is undoubtedly the parotidectomy. Parotid gland tumors are among the most common neoplasms in the head and neck region, and a variable portion (Linder TE et al., 1997; Bussu F et al., 2011; May JS, 1989). Ranging from 17% up to 100% of patients who underwent parotidectomy are affected by Frey's syndrome, depending whether or not they performed specific test. Grossly half of them notice symptoms and feel the gustatory sweating. Around 13-23% of patients consider their symptoms troublesome and severe (Laskawi RT et al., 1996; May JS, 1989). Potential negative social and psychologic implications of this condition can be significant, and treatment ranging from topical agents (glycopyrrolate) to local injections of botulinum toxin (Botox) to surgical intervention (i.e. temporoparietal fascia flap interposition) should be offered to patients (Hays LL, 1982). Moreover the Frey's syndrome, in addition to the gustatory sweating and flushing almost constant with a variable severity, can be associated with other atypical symptoms. The sensation of heat, itch and pain in the distribution of the auriculotemporal nerve were not mentioned as accompanying symptoms in the original description of the syndrome by Frey (Frey L., 1923). The pain is an uncommon finding, reported in less than 10% of cases (Bednarek J et al., 1976). It can be an early symptom and may remain the only one. Usually described as constant aching or burning, De Benedettis et al. (1990) reported two cases in which pain was the predominant symptom. Gustatory itch was described anecdotally by Ricks et al. (2010) as a sequela of superficial parotidectomy; a neurophysiological pathway involving acetylcoline and histamine has been proposed to explain this phenomenon. It cannot be ruled out that the presence of pain and itch is under-reported in the literature because they are generally not predominant, and the patient is often not specifically asked about. A systematic comprehensive assessment of Frey related complaints is currently missing. Most studies describe a single manifestation or the predominant ones basing simply on the absence or presence of symptoms and signs (Jansen S et al., 2017) without a graduation of them.

Study design and setting This will be a no-profit observational cross-sectional pilot study. Patients addressed to the Otolaryngology Unit of our Institution with a diagnosis of Frey syndrome will be consecutively enrolled, if matching inclusion criteria. The expected duration of the study will be two years.

Objectives

Primary

* To describe the prevalence of typical and atypical signs and symptoms of Frey's syndrome, the affected areas and the severity of each symptom/sign Secondary
* To describe the global severity of the Frey's syndrome in the group of the study;
* To describe the severity of Frey's syndrome in relation to the history data (etiology, age, sex, comorbidities, surgical procedure, age of onset)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Frey's syndrome

Exclusion Criteria:

* Patients already treated for Frey syndrome, with any therapy

  * History of radiation therapy of the head-neck district
  * Patients affected by neurologic diseases

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by Frey's syndrome after parotidectomy for parotid gland tumors
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
To describe the prevalence and the severity of typical and atypical signs and symptoms of Frey's syndrom | five years

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Raffaella Marchese, Roma, Italy

IPD SHARING:
Plan to Share IPD: No